CLINICAL TRIAL: NCT02426970
Title: Are Acceptance and Commitment Related to Treatment Response in Chronic Low Back Pain
Acronym: COP-PAIN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2014/AD-01; 2014-A01373-44 (Other: RCB number)
Record Dates: First submitted 2015-04-20; First posted 2015-04-27 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lumbar spine pain inpatients: The study population corresponds to inpatient rehabilitative care for lumbar spine pain in the Departments of Physical Medicine and Functional Rehabilitation at the Nîmes and Montpellier University Hospitals.

SUMMARY:
The main objective of this study is to evaluate whether acceptance (measured by the AAQ-II questionnaire) is prognostic of algo-functional changes measured by the Oswestry Disability Index, ODI) at 6 months.

DETAILED DESCRIPTION:
The secondary objectives are:

A. To search for correlations between the acceptance score (AAQ-II Questionnaire) and scores for coping (CSQ), avoidance (FABQ), understanding (BBQ), anxiety and depression (HADS) and quality of life (SF-12) at baseline.

B. To describe the kinetics of changes in various parameters (acceptance, coping, avoidance, understanding, anxiety and depression, quality of life, ODI) over 6 months.

C. To evaluate the agreement between two methods of questionnaire presentation: Paper collection versus collection by Tablet PC.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been informed about the study, and is not opposed to the study
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 6 month of follow-up
* The subject has chronic back pain that is not post-operative in nature and that has lasted for more than 3 months
* The subject accepts the re-education curriculum.

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to participate
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The subject has a history of chronic obstructive pulmonary disease, cardiovascular disease, rheumatoid arthritis, lupus, spondylitis or neoplastic disease.
* Patient currently under psychological treatment

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to inpatient rehabilitative care for lumbar spine pain in the Departments of Physical Medicine and Functional Rehabilitation at the Nîmes and Montpellier University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Classification of the patient as a responder or a non responder | 6 months
  The response to treatment will be evaluated by the ODI (Oswestry Disability Index) at 6 months: a patient will be considered as a responder when the absolute change between the score at 6 months and inclusion is at least 10 points (Ostelo RW et al., 2008).
  This outcome is a qualitative variable with two options: responder or non-responder. The fact that we define in an apriori fashion who is a responder or not does not mean that we have created multiple outcomes. This is a single outcome.
Acceptation and Action Questionnaire - II (AAQ-II) score | Day -7 (inclusion)

SECONDARY OUTCOMES:
the AAQ-II Score | Day 0
the AAQ-II Score | Month 1
the AAQ-II Score | Month 3
the AAQ-II Score | Month 6
Oswestry Disability Index | Day -7
Oswestry Disability Index | Day 0
Oswestry Disability Index | Month 1
Oswestry Disability Index | Month 3
Oswestry Disability Index | Month 6
Coping Strategies Questionnaire in French (CSQ-F) | Day -7
Coping Strategies Questionnaire in French (CSQ-F) | Day 0
Coping Strategies Questionnaire in French (CSQ-F) | Month 1
Coping Strategies Questionnaire in French (CSQ-F) | Month 3
Coping Strategies Questionnaire in French (CSQ-F) | Month 6
The Back Beliefs Questionnaire | Day -7
The Back Beliefs Questionnaire | Day 0
The Back Beliefs Questionnaire | Month 1
The Back Beliefs Questionnaire | Month 3
The Back Beliefs Questionnaire | Month 6
The Fear-Avoidance Beliefs Questionnaire | Day -7
The Fear-Avoidance Beliefs Questionnaire | Day 0
The Fear-Avoidance Beliefs Questionnaire | Month 1
The Fear-Avoidance Beliefs Questionnaire | Month 3
The Fear-Avoidance Beliefs Questionnaire | Month 6
The Hospital Anxiety and Depression Scale | Day -7
The Hospital Anxiety and Depression Scale | Day -0
The Hospital Anxiety and Depression Scale | Month 1
The Hospital Anxiety and Depression Scale | Month 3
The Hospital Anxiety and Depression Scale | Month 6
The SF-12 questionnaire | Day -7
The SF-12 questionnaire | Day 0
The SF-12 questionnaire | Month 1
The SF-12 questionnaire | Month 3
The SF-12 questionnaire | Month 6
Average pain over the last 8 days measured via visual analog scale. | Day -7
Average pain over the last 8 days measured via visual analog scale. | Day 0
Average pain over the last 8 days measured via visual analog scale. | Month 1
Average pain over the last 8 days measured via visual analog scale. | Month 3
Average pain over the last 8 days measured via visual analog scale. | Month 6
Maximum pain over the last 8 days measured via visual analog scale. | Day -7
Maximum pain over the last 8 days measured via visual analog scale. | Day 0
Maximum pain over the last 8 days measured via visual analog scale. | Month 1
Maximum pain over the last 8 days measured via visual analog scale. | Month 3
Maximum pain over the last 8 days measured via visual analog scale. | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes